CLINICAL TRIAL: NCT04072354
Title: A Randomized, Double-blind, Parallel-group, Placebo-controlled, Fixed-dose, Multicenter Study to Evaluate the Efficacy and Safety of SEP-363856 in Acutely Psychotic Subjects With Schizophrenia
Brief Title: A Clinical Trial to Study the Efficacy and Safety of an Investigational Drug in Acutely Psychotic People With Schizophrenia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Development & Commercialization, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SEP361-301; 2019-000470-36 (EudraCT Number)
Record Dates: First submitted 2019-08-26; First posted 2019-08-28 (Actual); Last update posted 2024-06-26 (Actual); Status verified 2024-06

CONDITIONS: Schizophrenia
Keywords: acute psychosis; schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — SEP-363856

STUDY DESIGN:
Intervention Model Description: randomized, double-blind, parallel-group, placebo controlled, fixed-dose multicenter study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: double-blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- SEP-363856 50mg (Experimental): SEP-363856 50mg dosed once daily
  Interventions: Drug: SEP-363856 50mg
- SEP-363856 75mg (Experimental): SEP-363856 75mg dosed once daily
  Interventions: Drug: SEP-363856 75mg
- Placebo (Placebo Comparator): Placebo dosed once daily
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SEP-363856 50mg — SEP-363856 50mg tablet dosed once daily
  Arms: SEP-363856 50mg
Drug: SEP-363856 75mg — SEP-363856 75mg tablet dosed once daily
  Arms: SEP-363856 75mg
Drug: Placebo — Placebo tablet dosed once daily
  Arms: Placebo

SUMMARY:
A clinical trial to study the efficacy and safety of an investigational drug in acutely psychotic people with schizophrenia. Participants in the study will either receive the drug being studied or a placebo. This study is accepting male and female participants between 13 years old -65 years old who have been diagnosed with schizophrenia. This study will be conducted in 70 locations worldwide. The study will last up to 9 weeks total time.

DETAILED DESCRIPTION:
This is a multicenter, randomized, double-blind, parallel-group, fixed-dosed study evaluating the efficacy and safety of two doses of SEP-363856 (50 and 75 mg/day) versus placebo over a 6-week Treatment Period in acutely psychotic subjects with schizophrenia. This study is projected to randomize approximately 435 subjects (18-65 years) to 3 treatment groups (SEP-363856 50 mg/day, SEP-363856 75 mg/day, or placebo) in a 1:1:1 ratio. In addition, the study will randomize approximately 90 adolescent subjects (13-17 years) in a 1:1:1 ratio to the 3 treatment groups (with approximately 30 subjects per group) in a separate cohort. Treatment assignment will be stratified by country. Study drug will be taken once a day and may be taken with or without food.

This study is designed to test the hypothesis that, treatment with SEP-363856 in adult subjects with schizophrenia will result in significantly greater reduction (i.e. improvement) in PANSS total score and CGI-S score at Week 6 from Baseline when compared to placebo. The overall Type I error is controlled for two hierarchical families of hypotheses. The first family includes hypotheses about the testing of change from Baseline in PANSS total score at Week 6 between each of the SEP-363856 dose levels vs. placebo. The second family of hypotheses are about the testing of change from Baseline in CGI-S score at Week 6 between each of the SEP-363856 dose levels vs. placebo.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subject between 13 to 65 years of age (inclusive) at the time of consent.
2. Subject or subjects parent/legal guardian [adolescents] must give written informed consent and privacy authorization prior to participate in the study; adolescents must also provide informed assent..
3. Subject meets DSM-5 criteria for schizophrenia as established by clinical interview at screening
4. Subject must have a CGI-S score ≥ 4
5. Subject must have a PANSS total score ≥ 80 and a PANSS item score ≥ 4 on 2 or more of the following PANSS items: delusions, conceptual disorganization, hallucinations, and unusual thought content
6. Subject has an acute exacerbation of psychotic symptoms (persisting no longer than 2 months prior to providing informed consent).
7. Subject has marked deterioration of functioning in one or more areas.
8. Subject is, in the opinion of the Investigator, generally healthy based on screening medical history, PE, neurological examination, vital signs, ECG, and clinical laboratory values.

Exclusion Criteria:

1. Subject has a DSM-5 diagnosis or presence of symptoms consistent with a DSM-5 diagnosis other than schizophrenia. Exclusionary disorders include but are not limited to alcohol use disorder (within past 12 months), substance (other than nicotine or caffeine) use disorder within past 12 months or lifetime history of significant substance abuse that in the opinion of the Investigator or Sponsor, may have had a significant and potentially permanent impact of the brain or other body systems, major depressive disorder, bipolar I or II disorder, schizoaffective disorder, obsessive compulsive disorder, and posttraumatic stress disorder. Symptoms of mild to moderate mood dysphoria or anxiety are allowed so long as these symptoms are not the primary focus of treatment.
2. Subject is at significant risk of harming self, others, or objects based on Investigator's judgment.
3. Subject has any clinically significant unstable medical condition or any clinically significant chronic disease that in the opinion of the Investigator, would limit the subject's ability to complete and/or participate in the study:
4. Female subject who is pregnant or lactating
5. Subject has any clinically significant abnormal laboratory value(s) at Screening as determined by the investigator.

Ages: 13 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 463 (Actual)
Dates: Start 2019-09-11 (Actual); Primary Completion 2023-05-12 (Actual); Study Completion 2023-09-12 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Positive and negative syndrome scale (PANSS) total score at Endpoint (Week 6) | Baseline and Week 6
  PANSS is comprised of 30 items and 3 subscales (Positive, Negative, General Psychopathology). An anchored Likert scale from 1 - 7, where values of 2 and above indicate the presence of progressively more severe symptoms, is used to score each item. Individual items are then summed to determine scores for the 3 subscales, as well as a total score. PANSS Positive subscale score range: 7-49. PANSS Negative subscale score range: 7-49. PANSS General Psychopathology subscale score range: 16-112. PANSS total score range: 30-210.

SECONDARY OUTCOMES:
Change from Baseline in Clinical Global Impressions - Severity (CGI-S) score at Endpoint (Week 6) | Baseline and Week 6
  The CGI-S is a single-item clinician-rated assessment of the subject's current illness state on a 7-point scale (score range: 1-7), where a higher score is associated with greater illness severity.

CONTACTS AND LOCATIONS:
Locations (57):
- United States (18):
  - Woodland International Research Group, LLC, Little Rock, Arkansas
  - Advanced Research Center, Inc., Anaheim, California
  - CITrials, Bellflower, California
  - Synergy San Diego, Lemon Grove, California
  - Alliance for Research, Long Beach, California
  - Catalina Research Institute, Montclair, California
  - California Neuropsychopharmacology Clinical Research Institute (CNRI-LA, LLC), Pico Rivera, California
  - UCSD Medical Center,UCSD Department of Psychiatry, San Diego, California
  - Larkin Behavioral Health Services, Hollywood, Florida
  - Research Centers of America, Hollywood, Florida
  - South Florida Research Phase I-IV, Inc., Miami Springs, Florida
  - Advanced Discovery Research LLC, Atlanta, Georgia
  - Atlantic Center for Medical Research, Atlanta, Georgia
  - iResearch Atlanta, LLC, Decatur, Georgia
  - CBH Health, LLC, Gaithersburg, Maryland
  - Precise Research Centers, Flowood, Mississippi
  - Midwest Clinical Research Center, Dayton, Ohio
  - Community Clinical Research, Austin, Texas
- Bulgaria (7):
  - State Psychiatric Hospital - Pazardzhik AD-Department of Active Treatment of Men Department for Active Treatment of Woman Department of Active Treatment of Mean and Woman, Pazardzhik
  - UMHAT-Dr. Georgi Stranski EAD-First Psychiatric clinic, Pleven
  - Mental Health Center-Sofia EOOD - Unit for Active Treatment of Persons with serious Mental Disorders, Sofia
  - UMHAT Alexandrovska EAD, First Department of Psychiatry at Clinic of Psychiatry, Sofia
  - UMHAT Alexandrovska EAD, Second Department of Pshychiatry at Clinic of Psychiatry, Sofia
  - Mental Health Center-Veliko Tarnovo EOOD-Deparmtentsof psychiatry for active treatment of persons with acute psychotic disorders, Veliko Tarnovo
  - Mental Health Center - Vratsa EOOD-Department of General Psychiatry, Vratsa
- Colombia (3):
  - E.S.E Hospital Mental de Antioquia - Unidad de Investigación, Bello, Antioquia
  - Centro de Investigaciones del Sistema Nervioso Limitada - Grupo CISNE Ltda, Bogotá
  - Centro de Investigaciones y Proyectos en Neurociencias CIPNA, Bogotá
- Russia (8):
  - State Budgetrary Institution of Healthcare Regional Clinical Specialized Psychiatric Hospital #1, Chelyabinsk
  - SBIH of Moscow "Psychiatric Clinical Hospital #4 n.a. P.B. Gannushkin", Moscow
  - State Budgetary Institution of Healthcare of nizhniy Novgorod region "Clinical Psychiatric Hosptial #1 of Nizhniy Novgorod, Nizniy Novgorod
  - State Budgetary Healthcare Institution of Republic Karelia "Republican Psyhiatric Hospital", Petrozavodsk
  - FSBI "NMRC of Psychiatry and Neurology named after V.M. Bekhterev" MoH RF, department 12, Saint Petersburg
  - FSBI 'NMRC of Psychiatry and Neurology named after V.M. Bekhterev MoH RF, department 12, Saint Petersburg
  - State Budgetary Institution of Healthcare "Samara Regional Clinical Psychiatric Hospital", Samara
  - State Institution of Healthcare Saratov City Clninical Hospital #2, named after V.I. Razumovskiy psychiatric deparmtents, Saratov
- Serbia (11):
  - Clinical Center "Dr. Dragisa Misovic-Dedinje" Clinic of Psychiatry, Belgrade
  - Clinical Center Nis, Center of Mental Health Protection, Belgrade
  - Institute of Mental Health, Belgrade
  - Special Hospital for Psychiartric Diseases Gornja Toponica, Stevana, Sindjelica 39, Gornja Toponica
  - Special Hospital for Psychiatric Diseases "Kovin",, Kovin
  - Special Neuropsychiatric Hospital Kovin, Kovin
  - Clinical Center Kragujevac, Clinic of Psychiatry, Kragujevac
  - University Clinical Center Nis, Clinic of Psychiatry, Niš
  - Special Hospital for Psychiatric Diseases "SVeti Vracevi",, Novi Kneževac
  - Clinical Center of Vojvodina, Clinic of Psychiatry, Novi Sad
  - Special Hospital for Psychiatric Diseases, Vršac
- Ukraine (10):
  - 15, Medychna St, Ivano-Frankivsk
  - 2-A Metalurgiv st, Kropyvnytskyi
  - Dr. Vladyslav Demchenko, Kyiv
  - 103 Kyrylivska St, Kyiv
  - Communal Noncommercial Enterprise of Lviv Regional Council Lviv Regional Clinical Psychiatric Hospital, Department #25, Lviv
  - 9 Academician Vorobiov St, Odesa
  - 1, Tsentraina Square, Oleksandrivka village, Lyman Region, Odesa Region, Odesa
  - 1 Medychna St, Poltava
  - Communal Non-commercial Enterprise Cherkasy Regional Psychiatric Hospital of Cherkasy Regional Council, Female Department #11, Male Department #12, Smila
  - Comm. Institution O.I. Yushchenko Vinnytsia Reg. Psychoneurologoical Hospital, Vinnytsia

IPD SHARING:
Plan to Share IPD: Yes
Anonymized Individual participant data (IPD) that underlie the results of this study will be shared with researchers to achieve aims pre-specified in a methodologically sound research proposal. Small studies with less than 25 participants are excluded from data sharing.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be available after marketing approval in global markets, or beginning 1-3 years following article publication. There is no end date to the availability of the data.
Access Criteria: Otsuka will share data on the Vivli data sharing platform which can be found here: https://vivli.org/ourmember/Otsuka/
URL: http://clinical-trials.otsuka.com